CLINICAL TRIAL: NCT06233474
Title: A Phase 1/2a Randomized, Double-Blind Placebo-controlled Study of Intra-articular Allocetra in Knee Osteoarthritis
Brief Title: Study of Intra-articular Allocetra in Knee Osteoarthritis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Enlivex Therapeutics Ltd. (Industry)
Collaborators: Nordic Bioscience Clinical Development (NBCD) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENX-CL-05-001
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Run-in phase followed by randomization phase
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Safety run-in phase - Allocetra increasing dose (Other): An open-label dose escalation phase to characterize the safety and tolerability of Allocetra injections to the knee in different doses and select the Allocetra dose and regimen for the randomized phase.
  Interventions: Drug: Allocetra
- Randomization phase - Placebo. (Placebo Comparator): Three intra-articular injections of placebo into the index knee.
  Interventions: Other: Placebo
- Randomization phase - Allocetra (Experimental): Three intra-articular injections of Allocetra at a selected dose, into the index knee.
  Interventions: Drug: Allocetra

INTERVENTIONS:
Drug: Allocetra — Allocetra-OTS is a cell-based therapy consisting of non-HLA-matched allogeneic peripheral blood mononuclear cells, induced to an apoptotic stable state
  Arms: Randomization phase - Allocetra; Safety run-in phase - Allocetra increasing dose
Other: Placebo — The control used in this study will be placebo. Placebo solution containing all excipients except for the Allocetra cells.
  Arms: Randomization phase - Placebo.

SUMMARY:
This is a double blind, randomized,multi-center study to evaluate the safety and efficacy of intra-articular administration of Allocetra compared to placebo in patients with symptomatic knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis is a degenerative disease driven by physical breakdown of the joint cartilage, together with a chronic inflammation within the knee space. Over time, many patients will develop worsening pain in the joint and functional impairment, which may ultimately require knee replacement.

Allocetra is an immunomodulatory cell-based therapy consisting of allogeneic peripheral blood mononuclear cells that have been modified to be engulfed by macrophages and reprogram them into their homeostatic state.

This Phase 1/2a study is comprised of an open-label safety run-in stage to characterize safety and tolerability of repeated injections of Allocetra to a target knee , followed by a double-blind randomized stage to evaluate the safety and efficacy of Allocetra repeated injections to the target knee compared to placebo, in moderate to severe knee osteoarthritis patients. Patients in both stages will be followed for up to a year following last treatment. the last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45 - 80 years.
2. Chronic osteoarthritis of index knee with knee-related joint pain
3. Radiographic evidence of knee osteoarthritis of K-L Grade 2 or 3 in the index knee.
4. Knee pain assessed daily over a period of 7 days during the screening period and following wash-out of pain medications
5. Patients with chronic knee pain for at least 3 months who have failed to respond adequately to conventional therapy.
6. Willing to abstain from other intra-articular treatments and adhere to the protocol restrictions for concomitant medications and therapies during the study.
7. Women of childbearing potential and all men must agree to use 2 methods of an adequate contraception prior to study entry and for the duration of study participation through 4 weeks following IP administration.

Exclusion Criteria:

1. Wheelchair bound.
2. Immunosuppressive therapy
3. Any known current or prior tumor of the index knee.
4. Any known history or current intra-articular or osseous infection of the index knee.
5. Any evidence of clinically significant active infection
6. Any known history of inflammatory arthropathy or crystal-deposition arthropathy
7. Any known severe systemic cartilage and/or bone disorder, such as, but not limited to, chondrodysplasia, osteogenesis imperfecta.
8. Body Mass Index (BMI) >40.
9. Any major surgical cartilage treatment within 6 months
10. Any ligamentous repair or malalignment correction in the index knee within 6 months
11. Major injury to the index knee, such as torn ligament or severe sprain within 6 months
12. Clinically relevant knee instability of the index knee
13. Severe hip osteoarthritis ipsilateral to the index knee.
14. Clinically significant widespread pain syndromes, e.g., fibromyalgia, long COVID syndrome.
15. Known coagulopathy, or use of anticoagulation medication or antiaggregant medication;.
16. certain tumors, severe cardiac, respiratory or hematologic diseases as defined in the protocol

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events and Serious adverse events following Allocetra-OTS injection | 7 months following Day 0
  Number and severity of adverse events (AEs), serious adverse events (SAEs) and treatment disruptions/ discontinuations throughout the study from Day 0 and up to 6 months following the last injection

SECONDARY OUTCOMES:
Weekly average of knee pain. | 4 months and 7 months following Day 0.
  Evaluation of change from baseline in weekly average of knee pain as measured using NRS (Numeric Rating Scale ) assessed at 3 months and 6 months from last study treatment.
  Scores range from 0-10 points, with higher scores indicating greater pain intensity
Change from baseline in WOMAC total score. | 4 months, 7 months and 13 months following Day 0.
  Change from baseline in Western Ontario and McMaster Universities Arthritis Index (WOMAC) total score at 3 months, 6 months, and 12 months from last study treatment administration.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Change in quality of life- Euro Quality of Life-5-dimension (EQ-5D) questionnaire | 4 months, 7 months and 13 months following Day 0.
  Change from baseline in QoL as measured by Euro Quality of Life-5-dimension (EQ-5D) questionnaire at 6 months and at 12 months from last study treatment administration.

CONTACTS AND LOCATIONS:
Overall Officials: Lital Weinfeld-Bergman, Study Director — Senior Director of Clinical Operations
Locations (12):
- Denmark (3):
  - Sanos Clinic Nordjylland, Gandrup
  - Sanos Clinic Herlev, Herlev
  - Sanos Clinic Syddanmark, Vejle
- Israel (6):
  - Barzilai Medical Center, Ashkelon
  - Rambam Medical Center, Haifa
  - Hasharon Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Ichilov - Tel Aviv Sourasky Medical Center, Tel Aviv
- Moldova (3):
  - IMSP Institutul de Cardiologie, Chisinau
  - Spitalul Clininc Republican "T. Mosneaga", Chisinau
  - IMSP Sptalul Clinic Municipal "Sfanta Treime", Chisinau